CLINICAL TRIAL: NCT07180927
Title: 4sCAR-DLL3 CAR-T Therapy Targeting Brain Tumors
Brief Title: DLL3 CAR-T Therapy Targeting Brain Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-25003
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma of Cerebellum
Keywords: CAR-T; Glioblastoma; DLL3
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR-DLL3 T Cell Therapy treating DLL3 positive glioblastoma (Experimental): Infusion of 4SCAR-DLL3 T cells at 10^6 cells/kg body weight via intravenous route
  Interventions: Biological: 4SCAR DLL3 T cells

INTERVENTIONS:
Biological: 4SCAR DLL3 T cells — Infusion of 4SCAR DLL3 T cells at 10^6 cells/kg body weight via intravenous route

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of Delta-like ligand 3 (DLL3)-specific CAR-T cell therapy in patients with DLL3 positive brain tumors including glioblastomas and diffused intrinsic pontine or midline gliomas (DIPG or DMG). Another goal of the study is to learn more about the function of the anti-DLL3 CAR-T cells and their persistency in patients.

DETAILED DESCRIPTION:
Glioblastoma (GBM) and other aggressive brain tumors remain among the most challenging cancers to treat, with limited therapeutic options and poor survival rates. GBM is known to express increased levels of certain antigens that can be targeted by T cells including chimeric antigen receptor-modified T (CAR-T) cells.

One promising target in this effort is DLL3, a protein highly expressed on the surface of certain tumor cells including GBM/DIPG/DMG and other central nervous system malignancies but with minimal presence in normal tissues. This expression pattern makes DLL3 an attractive target for precision CAR-T therapy treating brain tumors, which involves engineering a patient's own T cells to recognize and eliminate cancer cells expressing this specific marker.

This study aims to evaluate the safety, feasibility, and preliminary efficacy of DLL3-directed CAR-T cells in patients with recurrent or refractory brain tumors. These studies represent a critical step toward harnessing the immune system to fight traditionally treatment-resistant cancers, offering new hope for patients with few other options.

ELIGIBILITY:
Inclusion Criteria:

1. abilities to understand and the willingness to provide written informed consent;
2. patients are ≥ 2 and ≤ 70 years old;
3. recurrent or refractory brain tumor patients with measurable lesions. Patients have received standard care of medication, such as gross total resection with concurrent radio-chemotherapy (~54 - 60 Gy, TMZ). Patients must either not be receiving dexamethasone or receiving ≤ 4 mg/day at the time of leukopheresis;
4. Karnofsky performance score (KPS) ≥ 60;
5. life expectancy >3 months;
6. satisfactory bone marrow, liver and kidney functions as defined by the following: absolute neutrophile count ≥ 1500/mm^3; hemoglobin > 10 g/dL; platelets > 100000 /mm^3; Bilirubin < 1.5×ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5×ULN; creatinine < 1.5×ULN;
7. peripheral blood absolute lymphocyte count must be above 0.8×10^9/L;
8. satisfactory heart functions;
9. patients must be willing to follow the instructions of doctors;
10. women of reproductive potential (between 15 and 49 years old) must have a negative pregnancy test within 7 days of study start. Male and female patients of reproductive potential must agree to use birth control during the study and 3 months post study.

Exclusion Criteria:

1. a prior history of gliadel implantation 4 weeks before this study start or currently receiving antibody based therapies;
2. HIV positive;
3. tuberculosis infection not under control;
4. history of autoimmune disease, or other diseases require long-term administration of steroids or immunosuppressive therapies;
5. history of allergic disease, or allergy to immune cells or study product excipients;
6. patients already actively enrolled in other immune cell clinical study; patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 6 months
  Determine the toxicity profile the 4SCAR DLL3 cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Objective responses (complete response (CR) are assessed by the Response Evaluation Criteria in Glioblastoma (RECIST) v1.1 criteria.
Anti-tumor effects | 1 year
  Objective responses partial response (PR)) are assessed by the Response Evaluation Criteria in Glioblastoma (RECIST) v1.1 criteria.
The expansion of 4SCAR DLL3 T cells | 1 year
  Scale of CAR copies for efficacy
The persistence of 4SCAR DLL3 T cells | 1 year
  Scale of tumor burden for efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immuno Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No